CLINICAL TRIAL: NCT03609346
Title: Asian Registry of the BioFreedom™ BA9™ Drug-Coated Coronary Stent for Patients With ST Elevation Myocardial Infarction (STEMI) Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: Asian Registry of the BioFreedom Stent for STEMI Patients
Status: Completed | Type: Observational
Sponsor: Biosensors Europe SA (Industry)
Collaborators: Biosensors Interventional Technologies Pte Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-APAC-01
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
Keywords: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI: Arm: STEMI Intervention: PCI with 1 or more BioFreedom stents in patients presenting with a STEMI. Medication according to hospital practice.
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — The placement of 1 or more stents in the diseased coronary artery lesion(s).
  Other Names: Revascularization

SUMMARY:
The BioFreedom BA9 (Stainless Steel) Drug Coated Stent is an approved stent that is already commercially available in Europe and Asia. The purpose of this registry is to assess the safety and efficacy of the BioFreedom stent for treatment of a specific group of patients; patients with a myocardial infarction (STEMI). The objective is to capture patients' outcomes and antithrombotic strategies data using one or several BioFreedom Stents in the routine treatment of these STEMI patients.

DETAILED DESCRIPTION:
The purpose of this registry is to assess the safety and efficacy of the BioFreedom stent for treatment of STEMI patients. The objective is to capture patients' outcomes and antithrombotic strategies data using one or several BioFreedom Stents in the routine treatment of STEMI patients. This will be a fully observational post market registry designed to enroll 1000 STEMI patients at about 20 centers in up to 8 Asian countries where the BioFreedom BA9 (SS) DCS is available for clinical use.

The primary endpoint is LTF, which is a composite of cardiac death, target vessel-related reinfarction, and ischemia-driven target-lesion revascularization.

The investigators expect event rates of the composite of cardiac death, target vessel-related reinfarction, and ischemia-driven target-lesion revascularization to be 4.3% at one year as observed in the COMFORTABLE AMI study. Assuming a one-sided type I error (α) of 0.025, and a non-inferiority margin of 1.9%, a cohort of 1000 patients will have more than 80% power to conclude non-inferiority. The complete data analysis will be described in a Statistical Analysis Plan (SAP) that will be finalized and signed before the one year database lock.

Primary and secondary endpoint related events will be adjudicated by independent adjudicators. The study will be monitored per a monitoring plan, data will be collected in an electronic data capture system.

All enrolled patients will be followed up at 1, 4 and 12 months to collect information on their current status, review of cardiac medication taken and any adverse events that they have experienced.

Both CERC and Biosensors will follow company SOP's which are GCP and ISO 14155:2011 compliant.

ELIGIBILITY:
Inclusion Criteria:

1. STEMI patients treated with one or several BioFreedom stent(s) within 12h of symptom onset
2. Patients who agree to comply with the follow up requirements.
3. Patients with a life expectancy of > 1 year at time of consent.
4. Patients eligible to receive dual anti platelet therapy (DAPT). The establishment of the DAPT regimen is at the physician's discretion.

Exclusion Criteria:

1. Patients in cardiogenic shock
2. Any out of hospital cardiac arrest
3. Glasgow score < 15
4. Patients unable or unwilling to give documented informed consent
5. Patients with any PCI 6 months prior to the baseline procedure
6. Patients taking part in another interventional trial which has not completed follow-up for the primary endpoint
7. Patient has received an additional stent different from a BioFreedomBA9 (SS) DCS stent during the index procedure.
8. Pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry is open to all patients presenting with STEMI and treated with one or more BioFreedom BA9 (SS) DCS.
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 12 months
  TLF (Target Lesion Failure) defined as composite of cardiovascular death, target-vessel related myocardial infarction (Q-wave and non-Q-wave), or ischemia-driven target lesion revascularization within 12 months (device-oriented outcome per ARC2 definitions).

SECONDARY OUTCOMES:
1. All-cause mortality | 12 months
  1. All-cause mortality
2. Cardiovascular death | 12 months
  2. Cardiovascular death (cardiovascular and undetermined)
3. The composite of cardiac death, Target Lesion (TL)-related myocardial infarction and TL-related definite or probable stent thrombosis | 12 months
  3. The composite of cardiac death, Target Lesion (TL)-related myocardial infarction and TL-related definite or probable stent thrombosis at one year
4. Stroke disabling and non-disabling ARC definition | 12 months
  4. Stroke disabling and non-disabling ARC definition
5. Myocardial infarction (according to the Third Universal Definition) a. Q wave, non-Q wave and all myocardial infarctions | 12 months
  5. Myocardial infarction (according to the Third Universal Definition)
  a. Q wave, non-Q wave and all myocardial infarctions
6. ARC2 ST | 12 months
  6. ARC2 ST
7. Clinically driven TLR at any follow-up time point | 12 months
  7. Clinically driven TLR at any follow-up time point
8. Clinically driven target vessel revascularization | 12 months
  8. Clinically driven target vessel revascularization
9. Any revascularization within 12 months following the index procedure, unless they are planned within the 1st month | 12 months
  9. Any revascularization within 12 months following the index procedure, unless they are planned within the 1st month
10. Bleeding per BARC criteria a. BARC 3 to 5 | 12 months
  10. Bleeding per BARC criteria
  a. BARC 3 to 5

CONTACTS AND LOCATIONS:
Locations (5):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Tan Tock Seng Hospital, Singapore, Singapore
- Seoul National University Bundang Hospital, Seoul, South Korea
- Mackay Memorial Hospital, Taipei, Taiwan
- Her Majesty Cardiac Centre, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong PJL, Chui SF, Tam FC, Nguyen QT, Tsai CT, Kang WC, Nuruddin AA, Singh R, Chotinaiwattarakul C, Lee M. Polymer free biolimus coated stents to treat acute ST-elevation myocardial infarction in Asian patients. Catheter Cardiovasc Interv. 2024 Dec;104(7):1406-1413. doi: 10.1002/ccd.31263. Epub 2024 Oct 21. PMID 39434554